CLINICAL TRIAL: NCT02620670
Title: Evaluation of the Effect of Moderate-intensity Physical Activity on Glycemic Variability in Individuals With Visceral Obesity and Normal Weight Without Changes in Glucose Tolerance
Brief Title: Evaluation of the Effect of Moderate-intensity Physical Activity on Glycemic Variability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Esperanza Martínez-Abundis, PhD. Esperanza Martínez-Abundis, University of Guadalajara
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EAFVG
Record Dates: First submitted 2015-09-10; First posted 2015-12-03 (Estimated); Last update posted 2018-04-30 (Actual); Status verified 2018-01

CONDITIONS: Obesity
Keywords: Physical Activity; Glycemic Variability
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Individuals with obesity (Active Comparator): Body mass index (BMI) is 30.0 to 39.9 kg / m2 and a waist circumference greater than 80 cm in women and 90 cm for men Physical activity of moderate intensity for 3 days
  Interventions: Behavioral: Physical activity of moderate intensity for 3 days
- Individuals with normal weight (Active Comparator): Body mass index BMI is 18.5 to 24.9 kg / m2 with lower waist circumference of 80 cm for women and 90 cm for men Physical activity of moderate intensity for 3 days
  Interventions: Behavioral: Physical activity of moderate intensity for 3 days

INTERVENTIONS:
Behavioral: Physical activity of moderate intensity for 3 days — The intervencion consist in a moderate-intensity physical activity exercise is a heart rate between 60 and 70% of maximum heart beats per minute for at least 30 minutes for three days

SUMMARY:
Obesity is a major public health problem on the world and Mexico too, in addition the obesity develops chronic non-communicable diseases (NCD) such as type 2 diabetes mellitus (T2DM) and cardiovascular disease (CVD). So the phenomenon of obesity is studied in many investigations to know their causes, prevention and treatment.

Participation of body fat and especially in the visceral area is well documented in the appearance of T2DM; however, it is quite interesting that found that not all individuals with visceral obesity have impaired glucose tolerance, prediabetes or T2DM; but they are presented as normoglycemic individuals with obesity.

Currently, it is recognized that physical activity influences the concentrations of plasma glucose, and promoting their utilization in peripheral tissues, to be used as an energy source, through the regulation of glucose transporters in tissues such as the muscle, so might influence the glycemic variability, and therefore is of interest to this study to evaluate the effect of physical activity of moderate intensity on the glycemic variability of individuals with visceral obesity and normal weight without alterations in tolerance glucose.

DETAILED DESCRIPTION:
A quasi-experimental longitudinal and analytical study, consisting of two groups were carried out: a group of individuals with visceral obesity and other individuals with normal weight; both groups with no alteration in glucose tolerance. The world of work will be patients 30-40 years of age; for the group of individuals with visceral obesity body mass index (BMI) 30.0-39.9 kg/m2 and a waist circumference greater than 80 cm in women and 90 cm for men, and for the group of individuals with normal weight BMI 18.5-24.9 kg/m2 with lower waist circumference of 80 cm for women and 90 cm for men.

It will be confirmed by a curve oral glucose tolerance, that individuals do not have impaired glucose tolerance at baseline; likewise, they are determined serum levels of urea, creatinine, glutamic oxaloacetic transaminase (GOT), glutamic pyruvic transaminase (SGPT) and lipid levels (total cholesterol, triglycerides [TG], high-density lipoprotein cholesterol [HDL-C], low-density lipoprotein cholesterol [LDL-C] and very low density lipoprotein [VLDL]). BMI, waist circumference and body weight distribution (body fat percentage, visceral fat level, weight, lean body mass and percentage of water): On the other hand, at the beginning and end of the study the following determinations were obtained.

The study will last for 6 days. To measure glycemic variability on the first day they place a system of continuous glucose payment (MCG) through the iPro ™ 2 system (Medtronic MiniMed, Northridge) which determine interstitial glucose levels every five minutes. During the first 3 days the individual volunteer perform their usual activities, and three days later made moderate intensity physical activity for 30 minutes in the morning with fasting for 8-12 hours.

From the data obtained from MCG the mean amplitude of glucose excursions (MAGE), which will assess glycemic variability and area under the curve (AUC) was calculated. For statistical analysis, the Mann-Whitney U test, Fisher's exact test, Wilcoxon and linear regression was used. It is considered significant difference for p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Gender: male and female.
* Age: 30-40 years.
* Diagnosis of obesity and normal weight according to WHO:

Individuals with normal weight or BMI ≥ 18.5 to 24.9 kg / m2. Individuals with obesity or BMI ≥ 30 to 39.9 kg / m2.

• Diagnosis absence of visceral obesity according to WHO: Normal Weight; waist circumference: Women <80 cm and men <90 cm.

• Diagnosis of visceral obesity according to WHO: waist circumference: Women and men ≥ 80 cm ≥ 90 cm.

* What are sedentary during the past three months. Individuals committed in 15-30 minutes of physical activity exclusively by at least 3 times a week at most.
* No change in the oral glucose tolerance according to the ADA:

or fasting glucose <100 mg / dL and afterload glucose <140 mg / dL.

• written informed consent.

Exclusion Criteria:

* Women pregnant or lactating.
* Diagnosis of DM according to the ADA. Fasting glucose: ≥ 126 mg / dL glucose and afterload: ≥ 140 mg / dL.
* Thyroid disease and / or hypertension.
* Diagnosis of metabolic syndrome.
* Consumption of oral agents or other medicines and supplements with proven properties that modify the behavior of glucose.
* Liver enzymes: GOT and GPT concentrations twice normal.
* Changes in GFR according to the Cockcroft and Gault, with levels below 60 mL / min / 1.73 m2, which is suggestive of chronic kidney disease.
* Changes in serum lipid levels:

Total cholesterol <200 mg / dL Triglycerides <150 mg / dL HDL-C > 60 mg / dL or LDL-C <130 mg / dL

Ages: 30 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2015-04-15 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-12-27 (Actual)

PRIMARY OUTCOMES:
Mean amplitude of glucose excusions (MAGE) | 6 days
  Before and after the physical activity of moderate intensity outpatient daily glucose monitor iPro ™ 2

SECONDARY OUTCOMES:
Body mass index | 6 days
  Before and after the physical activity of moderate intensity
Waist circumference | 6 days
  Before and after the physical activity of moderate intensity
Postprandial glucose | 6 days
  Before and after the physical activity of moderate intensity outpatient daily glucose monitor iPro ™ 2

CONTACTS AND LOCATIONS:
Overall Officials: Esperanza Martínez-Abundis, PhD, Principal Investigator — Institute of Experimental and Clinical Therapeutics (INTEC), CUCS, University of Guadalajara
Locations (1):
- Institute of Experimental and Clinical Therapeutics (INTEC), CUCS, University of Guadalajara, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Undecided